CLINICAL TRIAL: NCT00098891
Title: A Phase I Study of an Oral Histone Deacetylase Inhibitor, MS-275 (NSC 706995, IND 61,198), in Combination With 13-Cis-Retinoic Acid in Metastatic Progressive Cancer.
Brief Title: MS-275 and Isotretinoin in Treating Patients With Metastatic or Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02634; JHOC-J0438; U01CA070095 (NIH); CDR0000396776 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Primary Central Nervous System Non-Hodgkin Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — entinostat; Isotretinoin

ARMS (1):
- Treatment (entinostat, isotretinoin) (Experimental): Patients receive oral MS-275 once on days 1, 8, and 15 and oral isotretinoin twice daily on days 1-21. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: entinostat; Drug: isotretinoin

INTERVENTIONS:
Drug: entinostat — Given orally
  Other Names: HDAC inhibitor SNDX-275; SNDX-275
Drug: isotretinoin — Given orally
  Other Names: 13-CRA; Amnesteem; Cistane; Claravis; Sotret

SUMMARY:
Phase I trial to study the effectiveness of combining MS-275 with isotretinoin in treating patients who have metastatic or advanced solid tumors or lymphomas. MS-275 may stop the growth of cancer cells by blocking the enzymes necessary for their growth. Isotretinoin may help cancer cells develop into normal cells. MS-275 may increase the effectiveness of isotretinoin by making cancer cells more sensitive to the drug. MS-275 and isotretinoin may also stop the growth of solid tumors or lymphomas by stopping blood flow to the cancer. Combining MS-275 with isotretinoin may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose-limiting toxicity and maximum tolerated dose of MS-275 when administered with isotretinoin in patients with metastatic, progressive, refractory, or unresectable solid tumors or lymphomas.

SECONDARY OBJECTIVES:

I. Determine, preliminarily, tumor response in patients treated with this regimen.

II. Determine the pharmacokinetic profile of this regimen in these patients.

OUTLINE: This is an open-label, dose-escalation study of MS-275.

Patients receive oral MS-275 once on days 1, 8, and 15 and oral isotretinoin twice daily on days 1-21. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of MS-275 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 12 patients are treated at the MTD.

Patients are followed monthly.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor or lymphoma

  * Metastatic, progressive, refractory, or unresectable disease
  * Not amenable to standard curative measures
* No known brain metastases
* Performance status - ECOG 0-2
* More than 3 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,000/mm^3
* Hemoglobin > 9 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* No suspected Gilbert's syndrome
* Creatinine ≤ 1.5 times ULN
* Creatinine clearance ≥ 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No unstable cardiac arryhthmia
* Able to take and retain oral medications
* No malabsorption problems
* No acute or chronic gastrointestinal condition
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception 1 month before, during, and 3 months after study treatment
* No known HIV positivity
* No weight loss > 10% within the past 2 months
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to MS-275 or isotretinoin
* No other uncontrolled illness
* No ongoing or active infection
* No seizure disorder
* No psychiatric illness or social situation that would preclude study participation
* More than 4 weeks since prior anticancer vaccine therapy
* More than 4 weeks since prior anticancer immunotherapy
* No concurrent anticancer vaccine therapy
* No concurrent anticancer immunotherapy
* More than 4 weeks since prior anticancer chemotherapy (6 weeks for nitrosoureas, mitomycin, or other agents known to cause prolonged marrow supression)
* No concurrent anticancer chemotherapy
* More than 4 weeks since prior anticancer hormonal therapy except gonadotropin-releasing hormone (GnRH) agonist therapy for non-castrated patients with prostate cancer
* Concurrent GnRH agonist therapy for non-castrated patients with prostate cancer allowed
* Concurrent luteinizing hormone-releasing hormone agonist therapy allowed provided there is evidence of tumor progression
* Concurrent adrenal steroid replacement therapy allowed
* No concurrent ketoconazole as second-line hormonal treatment for prostate cancer
* No concurrent corticosteroids except for treatment of refractory nausea or vomiting
* No other concurrent anticancer hormonal therapy
* More than 4 weeks since prior anticancer radiotherapy
* More than 2 weeks since prior palliative radiotherapy
* No concurrent anticancer radiotherapy
* More than 4 weeks since prior major surgery
* Recovered from all prior therapy
* No prior MS-275
* No prior oral isotretinoin

  * Isotretinoin for the treatment of acne allowed provided > 3 years since prior administration
* More than 4 weeks since other prior anticancer therapy
* No concurrent tetracycline
* No concurrent high-dose vitamin A
* No concurrent valproic acid
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-10; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities defined as an adverse event which is likely related to the study medication | 28 days
  Graded using the CTCAE version 3.0.
Maximum tolerated dose of entinostat and isotretinoin in combination | 28 days

SECONDARY OUTCOMES:
Pharmacokinetics | Up to day 21 of course 2
Adverse events defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment | Up to 30 days after completion of study treatment
  Graded using the CTCAE version 3.0. Summarized by dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pili, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States